CLINICAL TRIAL: NCT00038454
Title: A Phase II, Randomized, Single-Blind, Controlled Clinical Trial to Evaluate the Efficacy and Safety of Hemolink[Tm] (o-Raffinose Cross-Linked Human Hemoglobin) in Subjects Undergoing Primary Coronary Artery Bypass Grafting Surgery
Brief Title: Phase II Study To Evaluate The Safety and Efficacy of Hemoglobin Raffimer in Patients Undergoing First Time CABG Surgery
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hemosol (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HLK-213
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Cardiovascular Disease
Keywords: Oxygen Therapeutics; CABG; Transfusion
MeSH Terms: conditions — Cardiovascular Diseases | interventions — O-raffinose cross-linked human hemoglobin

INTERVENTIONS:
Drug: Hemolink (hemoglobin raffimer IV solution)

SUMMARY:
To evaluate the efficacy of Hemolink™ in combination with Intraoperative Autologous Donation (IAD) versus control (IAD alone) in facilitating avoidance of allogeneic RBC transfusion during and following primary CABG surgery

DETAILED DESCRIPTION:
All subjects who consent to take part in the protocol and who meet the inclusion/exclusion criteria will undergo the IAD harvest following a post-induction IAD harvest calculation. IAD blood will be collected into citrate-phosphate-dextrose-adenine 1 (CPDA-1) blood bags. All subjects will receive a volume of Hespan® equal to the volume of their IAD harvest (to a maximum of 1 liter) performed as a result of the harvest calculation (0-1200 mL inclusive). Additional volume replacement required owing to IAD >1000mL will be performed with crystalloid, as required. Subjects will be randomized into one of two treatment arms (Hemolink™ arm or control arm) upon meeting a transfusion trigger for the first time while on CPB. Randomization will be administered centrally. Subjects will be transfused upon reaching predetermined transfusion triggers, reflecting a decrease in hemoglobin concentration and/or oxygenation:

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria are eligible for inclusion in the study:

* Written Informed Consent.
* Age 18 through 80 years, inclusive.
* Scheduled for primary CABG surgery with CPB and are candidates for IAD.
* Post-induction hemoglobin, which will allow collection of 0-1200 mL inclusive of IAD blood to achieve a target hemoglobin of 7.5 g/dL at 15 minutes on-CPB.
* For women of childbearing potential only, able to use and using a highly-effective contraceptive method from the time of study screening through week 4 - 8 post CABG surgery (follow-up visit).

Note: International Conference on Harmonization (ICH) guidelines define a highly-effective contraceptive method as one with a failure rate of less than one percent when used consistently and correctly

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

* Previous treatment with Hemolink(tm) or any other hemoglobin-based oxygen carrier.
* Participation in any clinical trial of an investigational drug, device, or medical procedure within the two months prior to enrollment, or concurrent with participation in this study.
* History of stroke with residual paralysis or of transient ischemic attacks within 6 months prior to surgery.
* Congenital coagulation disorder or treatment with Coumadin within seven days prior to surgery.
* Alcohol or drug use within the 12 months prior to enrollment, which the investigator considers abusive.
* Planned simultaneous surgery (e.g., valve repair or carotid endarterectomy).
* Emergency CABG.
* Previous surgery using sternotomy.
* Current pregnancy or nursing.
* Chronic pancreatitis with or without pancreatic insufficiency.

Any subject who is medically cleared for both the surgical procedure and the intraoperative autologous donation will be eligible for enrollment in the study.

Medical clearance requires the following:

* No current congestive heart failure, New York Heart Association class IV.
* Most recent (within 1 year of surgery) ejection fraction must not be less than or equal to 25 percent, or left ventricular function of grade 4.
* No current uncontrolled hypertension.
* No current severe pulmonary disease which will render the subject at high risk of requiring prolonged post-operative ventilation.
* No serum creatinine > 2.0 mg/dL (177 umol/L).
* No known AST and ALT and bilirubin > 3 times the upper limit of normal.
* No uncontrolled angina within 24 hours prior to surgery despite maximal medical treatment, and/or presence of an intraaortic balloon pump preoperatively.
* No history of transmural myocardial infarction within the five days prior to the scheduled CABG surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180

CONTACTS AND LOCATIONS:
Locations (28):
- United States (19):
  - Kaiser Permanente Medical Center - San Francisco-Division of Cardiovascular Anesthesia, San Francisco, California
  - Stanford University Medical Center: Department of Anesthesiology, Stanford, California
  - Clinical Research Center, Sarasota, Florida
  - Heart and Vascular Care, Des Moines, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Englewood Hospital, Englewood, New Jersey
  - Robert Wood Johnson Hospital, New Brunswick, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina: Department of Anesthesiology, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Department of Anesthesiology, Columbus, Ohio
  - Veterans Affairs Medical Center, Portland, Oregon
  - Legacy Research, Portland, Oregon
  - UPMC Health System, Pittsburgh, Pennsylvania
  - Cardiovascular Anesthesia Research:Texas Heart Institute, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Medical College of Virginia: Department of Anesthesiology, Richmond, Virginia
- Canada (7):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Paul's Hospital/ Vancouver General Hospital, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Toronto Hospital - General Division, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Hopital Laval, Ste Foy, Quebec
- United Kingdom (2):
  - St. Thomas Hospital: Department of Anesthesia, London, England
  - Southampton General Hospital, Southampton, England

REFERENCES:
- [Background] Jahr JS, Lurie F, Driessen B, Davis JA, Gosselin R, Gunther RA. The HemoCue, a point of care B-hemoglobin photometer, measures hemoglobin concentrations accurately when mixed in vitro with canine plasma and three hemoglobin-based oxygen carriers (HBOC). Can J Anaesth. 2002 Mar;49(3):243-8. doi: 10.1007/BF03020522. PMID 11861341
- [Background] Kingma JG Jr, Sandhu R, Hamelin ND, Gendron D, Trudel Y, Bosa M, Stewart R, Fargey MB, Biro GP. The effects of hemodilution with Hemolink upon hemodynamics and blood flow distribution in anesthetized dogs. Artif Cells Blood Substit Immobil Biotechnol. 2001 Nov;29(6):465-81. doi: 10.1081/bio-100108551. PMID 11795632
- [Background] Topfer LA, Hailey D. Oxygen carriers ("blood substitutes"). Issues Emerg Health Technol. 2001 Jul;(21):1-6. PMID 11776287
- [Background] Scatena R, Giardina B. O-raffinose-polymerised haemoglobin. A biochemical and pharmacological profile of an oxygen carrier. Expert Opin Biol Ther. 2001 Jan;1(1):121-7. doi: 10.1517/14712598.1.1.121. PMID 11727541
- [Background] Cheng DC. Safety and efficacy of o-raffinose cross-linked human hemoglobin (Hemolink) in cardiac surgery. Can J Anaesth. 2001 Apr;48(4 Suppl):S41-8. PMID 11336436
- [Background] Caron A, Malfatti E, Aguejouf O, Faivre-Fiorina B, Menu P. Vasoconstrictive response of rat mesenteric arterioles following infusion of cross-linked, polymerized, and conjugated hemoglobin solutions. Artif Cells Blood Substit Immobil Biotechnol. 2001 Jan;29(1):19-30. doi: 10.1081/bio-100001253. PMID 11280681
- [Background] Toussaint M, Latger-Cannard V, Caron A, Lecompte T, Stoltz JF, Vigneron C, Menu P. Effects of three Hb-based oxygen-carrying solutions on neutrophil activation in vitro: quantitative measurement of the expression of adherence receptors. Transfusion. 2001 Feb;41(2):226-31. doi: 10.1046/j.1537-2995.2001.41020226.x. PMID 11239227
- [Background] Carmichael FJ, Ali AC, Campbell JA, Langlois SF, Biro GP, Willan AR, Pierce CH, Greenburg AG. A phase I study of oxidized raffinose cross-linked human hemoglobin. Crit Care Med. 2000 Jul;28(7):2283-92. doi: 10.1097/00003246-200007000-00017. PMID 10921554
- [Background] Cohn SM. Blood substitutes in surgery. Surgery. 2000 Jun;127(6):599-602. doi: 10.1067/msy.2000.106462. No abstract available. PMID 10840352
- [Background] Ning J, Wong LT, Christoff B, Carmichael FJ, Biro GP. Haemodynamic response following a 10% topload infusion of HemolinkTM in conscious, anaesthetized and treated spontaneously hypertensive rats. Transfus Med. 2000 Mar;10(1):13-22. doi: 10.1046/j.1365-3148.2000.00225.x. PMID 10760199
- [Background] Lieberthal W, Fuhro R, Andry C, Valeri CR. Effects of hemoglobin-based oxygen-carrying solutions in anesthetized rats with acute ischemic renal failure. J Lab Clin Med. 2000 Jan;135(1):73-81. doi: 10.1016/s0022-2143(00)70023-0. PMID 10638697
- [Background] Xue S, Paterson W, Valdez D, Miller D, Christoff B, Wong LT, Diamant NE. Effect of an o-raffinose cross-linked haemoglobin product on oesophageal and lower oesophageal sphincter motor function. Neurogastroenterol Motil. 1999 Dec;11(6):421-30. doi: 10.1046/j.1365-2982.1999.00171.x. PMID 10583849
- [Background] Freilich D, Branda R, Hacker M, Leach L, Barry B, Ferris S, Hebert J. Decreased lactic acidosis and anemia after transfusion of o-raffinose cross-linked and polymerized hemoglobin in severe murine malaria. Am J Trop Med Hyg. 1999 Feb;60(2):322-8. doi: 10.4269/ajtmh.1999.60.322. PMID 10072160
- [Background] Lieberthal W, Fuhro R, Freedman JE, Toolan G, Loscalzo J, Valeri CR. O-raffinose cross-linking markedly reduces systemic and renal vasoconstrictor effects of unmodified human hemoglobin. J Pharmacol Exp Ther. 1999 Mar;288(3):1278-87. PMID 10027869
- [Background] Glaser V. Fake blood market gets hemoglobin transfusion from reticulocytes. Nat Biotechnol. 1998 Aug;16(8):709. doi: 10.1038/nbt0898-709. No abstract available. PMID 9702757
- [Background] Macdonald RL, Zhang J, Weir B, Marton LS, Wollman R. Adenosine triphosphate causes vasospasm of the rat femoral artery. Neurosurgery. 1998 Apr;42(4):825-32; discussion 832-3. doi: 10.1097/00006123-199804000-00082. PMID 9574647
- [Background] Balion CM, Champagne PA, Ali AC. Evaluation of HemogloBind for removal of o-raffinose cross-linked hemoglobin (Hemolink) from serum. Clin Chem. 1997 Sep;43(9):1796-7. No abstract available. PMID 9299985
- [Background] Ali AC, Mihas CC, Campbell JA. Interferences of o-raffinose cross-linked hemoglobin in three methods for serum creatinine. Clin Chem. 1997 Sep;43(9):1738-43. PMID 9299969
- [Background] Kerger H, Tsai AG, Saltzman DJ, Winslow RM, Intaglietta M. Fluid resuscitation with O2 vs. non-O2 carriers after 2 h of hemorrhagic shock in conscious hamsters. Am J Physiol. 1997 Jan;272(1 Pt 2):H525-37. doi: 10.1152/ajpheart.1997.272.1.H525. PMID 9038975
- [Background] Baines AD, Christoff B, Wicks D, Wiffen D, Pliura D. Cross-linked hemoglobin increases fractional reabsorption and GFR in hypoxic isolated perfused rat kidneys. Am J Physiol. 1995 Nov;269(5 Pt 2):F628-36. doi: 10.1152/ajprenal.1995.269.5.F628. PMID 7503228
- [Background] Wong LT, Er SS, Ning J, Christoff B, Carmichael FJ. Hemolink-induced effects on intestinal motor function and attenuation of these effects by selected agents. Artif Cells Blood Substit Immobil Biotechnol. 1998 Nov;26(5-6):529-48. doi: 10.3109/10731199809117473. PMID 9844719
- [Background] Ali AC, Campbell JA. Interference of o-raffinose cross-linked hemoglobin with routine Hitachi 717 assays. Clin Chem. 1997 Sep;43(9):1794-6. No abstract available. PMID 9299984
- [Background] Arnoldo BD, Minei JP. Potential of hemoglobin-based oxygen carriers in trauma patients. Curr Opin Crit Care. 2001 Dec;7(6):431-6. doi: 10.1097/00075198-200112000-00010. PMID 11805546
- [Background] Caron A, Menu P, Faivre-Fiorina B, Labrude P, Alayash AI, Vigneron C. Cardiovascular and hemorheological effects of three modified human hemoglobin solutions in hemodiluted rabbits. J Appl Physiol (1985). 1999 Feb;86(2):541-8. doi: 10.1152/jappl.1999.86.2.541. PMID 9931189